CLINICAL TRIAL: NCT01142752
Title: Vaginal, Oral and Systemic Inflammation in Preterm Birth
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: KEK091/10
Record Dates: First submitted 2010-06-07; First posted 2010-06-11 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Local or Systemic Signs for Infection, Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, vaginal smears, oral specimens
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Control: Control group of women with uneventful pregnancy
- Population at risk with preterm birth: Women medically considered at risk for PTB and actually delivering preterm
- Population at risk without preterm birth: Women medically considered at risk for PTB but with uneventful pregnancy

SUMMARY:
The prevalence of preterm birth is not decreasing in the last decades despite of improving health care. Intrauterine infections are important in the etiology of preterm birth but the interconnection of systemic inflammation and preterm birth is not clear. Mechanisms of preterm birth should be assessed as preterm birth is the major risk factor for morbidity and mortality during birth, thus being important for the individual and regarding health costs.

No interventions will be carried out in this study.

Hypotheses:

1. There is a common etiology between oral and vaginal inflammation
2. Bacterial species are similar in vagina and oral cavity
3. There are similar oral and systemic immune reactions which provoke preterm birth
4. Inflammatory markers are found in pregnant women at risk and get back to normal post partum In this matched case control study of pregnant women local, systemic and oral inflammation markers and bacterial load are assessed to find out interconnections between these body compartments to allow for explanation of the etiology of preterm birth.

DETAILED DESCRIPTION:
Vaginal, oral and systemic inflammation in preterm birth

1. Summary

   The prevalence of preterm birth (PTB) is increasing. While intrauterine infections may be the primary cause of PTB, remote infections may also be part of the aetiology and risk for gestational complications. Predicting and identifying women at risk for delivering preterm is difficult. Comprehensive studies are needed to study all infectious and inflammatory processes that may be involved in birth complications. Social, ethnic and behavioural risks are part of the factors involved. Thus, case-control studies of infection in pregnancy must acknowledge and control for such other factors.

   The oral cavity provides a unique study model of periodontal infection and inflammation. Gingivitis and periodontitis have been associated with an elevated risk for PTB. A large entity of bacteria including both aerobic and anaerobic bacteria competent to elicit a systemic hyper-inflammatory host immune response can be identified in periodontal infection. Inflammation of the gingival tissues increases in pregnancy. Knowledge obtained through studies of clinical parameters as well as studies of bacteria and cytokines in oral, vaginal and blood samples in pregnant women at risk for preterm birth would establish evidence-based background for successful clinical strategies to prevent or reduce the risk for PTB.

   The objectives of the present matched case-control study of pregnant women are to investigate local and remote infection (microbiological analysis by culture, and DNA-DNA checkerboard) and inflammation (cytokine assays in samples from vaginal and oral samples), and routine clinical data in three groups of pregnant women:

   I. Women medically considered at risk for and WITH actual preterm birth delivery

   II. Women medically considered at risk for preterm birth delivery but who deliver WITHOUT birth complications

   III. Women with a normal uneventful pregnancy (control group)

   The investigators aim to test the following hypotheses regarding associations between oral infection and PTB:

   I. There is a shared infectious aetiology between oral and vaginal infections (primary outcome)

   II. In women at risk for PTB the vaginal and oral bacterial microbiota are similar

   III. There are similar systemic and/or local inflammatory responses (haematogenous dissemination and bacteraemia, feto-maternal immune response) that can be induced by vaginal and/or oral infection, contributing to PTB.

   IV. Elevated inflammatory markers are found at the onset of symptoms in pregnant women at risk for PTB and normalize after birth.
2. Current status in this field of research

   2.1. Introduction

   Preterm birth (PTB) is defined as delivery before 37 weeks of gestation and a birth weight of < 2500 grams. PTB is the most important determinant of perinatal morbidity and mortality. Among those born before 32 weeks of gestation many children will suffer from lifelong sequelae of prematurity ranging from mild to severe developmental disorders.
3. Detailed Research Plan

3.1. Scientific objectives (Aims)

The investigators aim to test the following hypotheses regarding associations between oral infection and PTB:

I. There is a shared infectious aetiology between oral and vaginal infections (primary outcome)

II. In women at risk for PTB the vaginal and oral bacterial microbiota are similar

III. There are similar systemic and/or local inflammatory responses (haematogenous dissemination and bacteraemia, feto-maternal immune response) that can be induced by vaginal and/or oral infection, contributing to PTB

IV. Elevated inflammatory markers are found at the onset of symptoms in pregnant women at risk for PTB and normalize after birth

3.2. Patient grouping

The study design is a longitudinal, non-interventional case-control study of pregnant women including (I) a control group of women with uneventful pregnancy

(II) a group of women medically considered at risk for PTB and actually delivering preterm

(III) a group of women medically considered at risk for PTB but with uneventful pregnancy.

Subjects will be examined at three time points (I) within 18-34 weeks of pregnancy when they get symptomatic

(II) within two days after delivery and

(III) 4-6 weeks post-partum. This would allow the investigators to compare all examined parameters between and within groups over the defined time frame.

Due to the medical inclusion criteria clinical medical/dental examinators cannot be blinded. At the first examination the clinicians will not know whether subjects belong to group II or group III. All laboratory processes will, however, be performed with no knowledge of group assignment.

The investigators intend to enrol a total of 180 pregnant women with a clinically perceived risk for PTB or at no/low risk based on routine clinical assessment criteria. Consecutive consenting pregnant women seeking care at, or are being referred to the Frauenspital, University of Berne will be asked to participate when admitted to the prenatal care unit because of risks for PTB, e.g. shortening of the cervical length, preterm contractions or prelabor premature rupture of membranes. The investigators anticipate a 10% dropout rate. They intend to continuously match subjects in the control group to those in the risk groups.

Consenting women will receive study examinations as well as obstetric standard of care during pregnancy provided by medical faculty investigators. Dental faculty investigators at the Department of Periodontology, University of Bern will perform dental examinations, data and sample collections from the participating subjects at either the Clinics of the Dental School or at the Frauenspital for bedridden pregnant women. There will be no specific dental interventions as part of the study. The dentists who normally provide care for study subjects will continue to do so. There are currently no known dental procedures that can reduce the risk for PTB. Dental procedures during pregnancy are considered at low or no risk to the pregnant women or the fetus.

The investigators will collect information on all medical and dental treatments performed during pregnancy. They will assess obstetric and dental clinical conditions, using procedures that they follow in both clinics. The investigators will also assess bacteria and fungi in vaginal and oral compartments, and serum and local vaginal/oral inflammatory markers (cytokines and C-reactive protein). They recognize that genetic and socio-economic factors as well as ethnicity are important factors in risks for PTB. The control group will therefore be paired and matched for gestational age, ethnicity, age, parity and smoking. The investigators anticipate that some of these subjects in the assigned no risk control group may actually deliver with PTB. Only women who deliver uneventfully will be included in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* Written informed consent

Exclusion Criteria:

* Matching with control patients not possible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women of more than 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2011-11; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Difference in systemic and local parameters of infection between patients at risk and controls | The study period is meant to be 2 years. Measures will be carried out during pregnancy, within 2 days after birth and 6 weeks post-partum.
  Oral, vaginal and placental infection parameters are measured during pregnancy, at birth and 6 weeks post partum. Samples are collected from blood, vaginal and placental (at birth) smears, histology, and oral smears. Measures include microbiologic culturing, gram stains, CRP, Cytokines (TNFalpha, IL-1beta, IL-6, IL-8, IL-10, PgE2). From blood samples a differential blood count, CRP, and cytokines are determined.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel V Surbek, Prof., Study Director — University women's hospital Bern
Locations (1):
- University Women's Hospital, Bern, Switzerland